CLINICAL TRIAL: NCT01956370
Title: Phase II - Evaluation of Safety and Efficacy of the PrePexTM Device for Rapid Scale up of Adult Male Circumcision Programs in Zimbabwe (Comparative Study)
Brief Title: Comparing the PrePex™ Device to Surgical MC for Rapid Scale Up of MC in Resource Limited Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ministry of Health and Child Welfare, Zimbabwe (Other)
Responsible Party: Principal Investigator, Prof. Mufuta Tshimanga, Public Health Physician, Department of Community Medicine, University of Zimbabwe, Ministry of Health and Child Welfare, Zimbabwe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MRCZ/A/1628 Comparative study
Record Dates: First submitted 2012-09-19; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: HIV
Keywords: Male Circumcision; HIV Prevention; Medical Device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PrePex™ device (Experimental): Intervention 'PrePex™ device for adult male circumcision
  Interventions: Device: PrePex™ device for adult male circumcision
- Surgical (Active Comparator): Adult male surgical circumcision
  Interventions: Procedure: Surgical circumcision

INTERVENTIONS:
Device: PrePex™ device for adult male circumcision — The PrePex™ device is designed to enable bloodless male circumcision procedure with no anesthesia and no sutures.
  Other Names: The PrePex Device; PrePex; PrePex™
  Arms: PrePex™ device
Procedure: Surgical circumcision — The penis will be surgically circumcised according to one of the WHO recommended circumcision methods as described in the Manual for Male Circumcision under Local Anaesthesia Version 2.5C January 2008
  Arms: Surgical

SUMMARY:
The protocol, approved by the Medical Research Council, was issued to assess the safety and efficacy of the non-surgical device for applying it to the national scale up of adult male circumcision in Zimbabwe

DETAILED DESCRIPTION:
Models show that to have the highest impact on the HIV epidemic, circumcision of up to 80% of men in high prevalence countries, where MC rates are low, needs to be achieved (UNAIDS 2009; Manicaland HIV/STD Prevention Project, 2008; Bollinger, et al, 2009). Hallett and colleagues in 2008 showed that for Zimbabwe specifically, HIV incidence could be reduced between 25% to 35% if about 50% of men are circumcised. All modelings conducted show that MC programs must be part of a comprehensive HIV prevention package as MC alone will not tip the HIV epidemic into a terminal decline.

The PrePex Device offers hope for rapid scale up of adult male circumcision in resource limited settings.

Once the safety and efficacy have been established, it is important to conduct operations research to determine how best to implement both device and surgical circumcisions in the national program. Thus, the Zimbabwe MOHCW is planning a three phase trial in order to determine the safety of the PrePexTM device, its performance and the ease of use in an implementation roll out.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 30 years
* Uncircumcised
* Wants to be circumcised
* Agrees to be circumcised by any of the study methods,PrePexTM or Surgical as appropriate
* HIV sero-negative
* Able to understand the study procedures and requirements
* Agrees to abstain from sexual intercourse and to keep caution not to directly rub the cut area if masturbating, for 8 weeks post removal (9 weeks total)
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision for a period of 8 weeks post removal (9 weeks total)
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study
* Subject agrees to anonymous video and photographs of the procedure and follow up visits
* Agrees to stay overnight at the Hospital in order to follow pain measurements in the first 16 hours

Exclusion Criteria:

* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* HIV sero-positive
* Subject with the following diseases/conditions: phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias, epispadias
* Known bleeding / coagulation abnormality
* Uncontrolled diabetes
* Subject that to the opinion of the investigator is not a good candidate
* Subject does not agree to anonymous video and photographs of the procedure and follow up visits
* Refusal to take HIV test.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Procedure time | 9 weeks
  To compare the total operative time of the PrePex Device circumcision procedure versus the total operative time of surgical circumcision procedure.

SECONDARY OUTCOMES:
Expectations of men regarding the procedure | 9 weeks
  Expectations of men regarding the procedure using questionnaires
Satisfaction rate of the procedure | 9 weeks
  Satisfaction with procedure using questionnaires and evaluations
Attitudes towards procedure | 9 weeks
  Attitudes towards procedure using questionnaires
Sharing information with family and friends | 9 weeks
  Sharing information with family and friends by evaluating weather subjects would recommend the procedure to others using questionnaires
Perception of norms | 9 weeks
  Perception of norms using questionnaires
Sexual relations, performance, satisfaction | 9 weeks
  Sexual relations, performance, satisfaction using questionnaires
Sexual behavior | 9 weeks
  Sexual behavior using questionnaires. Inquiring of sexual behavior before and after the circumcision, etc.
Sexual partner's attitudes | 9 weeks
  Sexual partner's attitudes using questionnaires and investigating the partner's behavior change as a result of her partner's circumcision.
Effect on daily activities | 9 weeks
  Effect on daily activities using questionnaires. Inquiring and finding out if the MC procedure caused any missing of working days.
Costs | 9 weeks
  Evaluating the cost of PrePex circumcision procedure when taking into account the following parameters:
  i. PrePex Procedure time and the resulting cost of provider's time ii. Cost of staff time for follow-up visits iii. Cost of equipment and supplies needed for the circumcision procedure
Cost-effectiveness | 9 weeks
  Cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gwinji, MBChB, MPH, Principal Investigator — PS- MoHCW
Locations (1):
- Znfpc Spilhaus Center, Harare, Zimbabwe

REFERENCES:
- [Derived] Hohlfeld A, Ebrahim S, Shaik MZ, Kredo T. Circumcision devices versus standard surgical techniques in adolescent and adult male circumcisions. Cochrane Database Syst Rev. 2021 Mar 31;3(3):CD012250. doi: 10.1002/14651858.CD012250.pub2. PMID 33786810
- [Derived] Tshimanga M, Mangwiro T, Mugurungi O, Xaba S, Murwira M, Kasprzyk D, Montano DE, Nyamukapa D, Tambashe B, Chatikobo P, Gundidza P, Gwinji G. A Phase II Randomized Controlled Trial Comparing Safety, Procedure Time, and Cost of the PrePex Device to Forceps Guided Surgical Circumcision in Zimbabwe. PLoS One. 2016 May 26;11(5):e0156220. doi: 10.1371/journal.pone.0156220. eCollection 2016. PMID 27227679
- See also: MRCZ — http://www.mrcz.org.zw/